CLINICAL TRIAL: NCT07043127
Title: Clinical Randomized Trial of the Influence of Rehabilitation Therapy Using Strength and Blood Flow Restriction Training on Muscular Fitness and Regeneration After Elective Hip Replacement
Brief Title: Impact of Rehabilitation Therapy Using Strength and Blood Flow Restriction Training on Muscular Fitness and Regeneration After Elective Hip Replacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B.Sc., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024_E
Record Dates: First submitted 2025-05-21; First posted 2025-06-29 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-05

CONDITIONS: Total Hip Arthroplasty (THA)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Regular Rehabilitation Training
  Interventions: Other: Sham-BFR
- Intervention Group (Experimental): BFR-Intervention during Rehabilitation Training
  Interventions: Other: BFR

INTERVENTIONS:
Other: Sham-BFR — The exercise protocol provides for units of approx. 25 minutes of BFR training five times a week as part of medical training therapy. Based on the initial strength measurements prior to rehabilitation, the training phase of the intervention group starts with 30% of the 1RM (calculated from the force-velocity profile) and 70% LOP in the operated leg and 75% of the 1RM (calculated from the force-velocity profile) in the unoperated leg. The patients are randomized into 2 groups: 1) intervention group, which receives a daily intervention with an occlusion pressure and the 2) control group, which receives a daily "Sham-BFR" intervention with an occlusion pressure of 20mmHg.
  Arms: Control Group
Other: BFR — The exercise protocol provides for units of approx. 25 minutes of BFR training five times a week as part of medical training therapy. Based on the initial strength measurements prior to rehabilitation, the training phase of the intervention group starts with 30% of the 1RM (calculated from the force-velocity profile) and 70% LOP in the operated leg and 75% of the 1RM (calculated from the force-velocity profile) in the unoperated leg. The patients are randomized into 2 groups: 1) intervention group, which receives a daily intervention with an occlusion pressure and the 2) control group, which receives a daily "Sham-BFR" intervention with an occlusion pressure of 20mmHg.
  Arms: Intervention Group

SUMMARY:
In the present project, the framework conditions of outpatient rehabilitation at the Bonn Center for Outpatient Rehabilitation will now be used to prove whether sports science-controlled strength and BFR training has a similar effect in the postoperative rehabilitation phase. Strength and BFR training in medical training therapy complements daily exercise therapy in order to ensure implementation in the guideline-based rehabilitation process. . The interventions are carried out as part of the exercise therapy units in outpatient rehabilitation ETM01 following the RTS hip and knee TEP basis KTL 2020.

ELIGIBILITY:
Inclusion Criteria:

* Ability for Rehabilitation
* Total Hip Arthroplasty Surgery during the last 4 Weeks

Exclusion Criteria:

* Sickle Cell Anemia
* Iatrogenic changes in the vessels of the lower Extremity (e.g. Stents)
* Open Wounds or Infections of the lower Extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength | Pre- (Baseline) to Post-Rehabilitation (after three weeks of outpatient rehabilitation)
  Muscle Strength will be assessed by isometric maximal contraction test on a leg press machine
Subjective Pain Level | Pre- (Baseline) to Post-Rehabilitation (after three weeks of outpatient rehabilitation)
  Visual analog scale (0-100mm)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No